CLINICAL TRIAL: NCT00627822
Title: Patient and Companion Perspectives on Medical Education in a Non-Teaching Private Hospital
Brief Title: Medical Education in a Private Hospital
Status: Completed | Type: Observational
Sponsor: Instituto do Cerebro de Brasilia (Other)
Responsible Party: Ricardo Afonso Teixeira MD PhD, Hospital Santa Luzia
Other Study IDs: HSL-EN
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Health Care Quality, Access, and Evaluation
Keywords: Medical students; Medical education; Private hospital; Patient satisfaction; Questionnaires
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ward: Patients in the hospital ward
- Emergency room: Patients in the emergency waiting room
- Intensive care unit: Family members of patients admitted to the intensive care unit

SUMMARY:
The purpose of this study is to assess patient and companion acceptability of medical education in a non-teaching private hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients in the hospital ward and in the emergency waiting room
* Family members of patients admitted to the intensive care unit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Private hospital: Patient and family members
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2005-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Patient and companion acceptability of medical education | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Teixeira, MD PhD, Study Director — Instituto do Cérebro de Brasília

REFERENCES:
- [Background] Benson J, Quince T, Hibble A, Fanshawe T, Emery J. Impact on patients of expanded, general practice based, student teaching: observational and qualitative study. BMJ. 2005 Jul 9;331(7508):89. doi: 10.1136/bmj.38492.599606.8F. Epub 2005 Jul 4. PMID 15996965
- [Background] O'Flynn N, Spencer J, Jones R. Consent and confidentiality in teaching in general practice: survey of patients' views on presence of students. BMJ. 1997 Nov 1;315(7116):1142. doi: 10.1136/bmj.315.7116.1142. No abstract available. PMID 9374890
- [Background] Grayson MS, Klein M, Lugo J, Visintainer P. Benefits and costs to community-based physicians teaching primary care to medical students. J Gen Intern Med. 1998 Jul;13(7):485-8. doi: 10.1046/j.1525-1497.1998.00139.x. PMID 9686716
- [Background] Cooke F, Galasko G, Ramrakha V, Richards D, Rose A, Watkins J. Medical students in general practice: how do patients feel? Br J Gen Pract. 1996 Jun;46(407):361-2. PMID 8983256
- [Background] Kupersmith J. Quality of care in teaching hospitals: a literature review. Acad Med. 2005 May;80(5):458-66. doi: 10.1097/00001888-200505000-00012. PMID 15851459